CLINICAL TRIAL: NCT01195194
Title: Pilot Study of Selection of Either Calcineurin Inhibitor(CNI)-Based or CNI-free Immunosuppressive Regimen Depending on the Result of Pre-transplantation Donor-specific T-cell Reactivity Measured by Enzyme-linked Immunosorbent Spot(ELISPOT) in Standard-risk Kidney Recipients.
Brief Title: Selection of Immunosuppression in Kidney Transplant Recipients Depending on Pre-transplant Donor-specific T-cell Reactivity.
Acronym: SIRES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Josep M Grinyo (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor-Investigator, Josep M Grinyo, Chief of the Nephrology Department- Hospital Universitari de Bellvitge, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIRES; 2007-002378-68 (EudraCT Number)
Record Dates: First submitted 2010-04-19; First posted 2010-09-06 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Disorder Related to Renal Transplantation
Keywords: T-cell lymphocyte allo-recognition; CNI-free immunosuppressive regimen; Enzyme-linked immunospot (ELISPOT)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A- negative pre-transplant ELISPOT (Experimental): Sirolimus: Start at 5 mg/day as soon as treatment allocation arrives to obtain targeting levels to 8 -15 ng/ml (immunoassay) in the first 3 months, followed by trough levels of 5-10 ng/ml.
  Interventions: Drug: PRE-TRANSPLANT (PRE=before)
- B- Positive pre-transplant ELISPOT (Experimental): Tacrolimus 0.1 mg/kg/12h starting as soon as treatment allocation arrives to obtain targeting troughs levels of 8-15 ng/ml the first 3 months, followed by trough levels of 5-10 ng/ml until the end of the study.
  Interventions: Drug: PRE-TRANSPLANT (PRE=before)

INTERVENTIONS:
Drug: PRE-TRANSPLANT (PRE=before) — All patients will start with Thymoglobulin 1 mg/kg before transplant followed by 0,5 mg/kg/d during the next 5 days (total accumulated 3,5 mg/kg).
  Steroids will be administered at 0,25 mg/kg/d until month 3rd, followed by 0,1 mg/kg/d thereafter.
  Mycophenolate Mofetil: Pre-transplant 2 grams iv. After transplantation 1g/12 hours, starting iv and changing to oral formulation as soon as patient starts with oral intake (targeting mycophenolic acid (MPA) C0h levels 2-5 µg/mL).

SUMMARY:
The objective is to assess if low pre-transplantation donor specific T-cell reactive patients measured by Enzyme-linked immunosorbent spot (ELISPOT)assay can be safely managed with Calcineurin inhibitor(CNI)-free Sirolimus(SRL)-based immunosuppression.

DETAILED DESCRIPTION:
Non randomized, pilot, prospective, open-label trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age of donor and recipient between 18 and 65 years.
2. End-stage renal disease and scheduled to receive a primary or secondary renal allograft from a cadaveric, a living-unrelated, or a living-related donor. Patients scheduled for a second transplant must have maintained their primary graft for at least 6 months after transplantation, with the exception of graft failure due to technical reasons.
3. Panel reactive antibody (PRA) ≤ 20%, with negative standard cross-match.
4. Women of childbearing potential must have a negative serum pregnancy test before randomization.
5. Women of childbearing potential must agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months following discontinuation of assigned treatment.
6. Signed and dated informed consent prior to transplantation.

Exclusion Criteria:

1. Multiple organ transplants
2. Recipients of adult or pediatric en bloc kidney transplants or dual transplantation or non-heart beating donors.
3. Evidence of active systemic or localized major infection.
4. Evidence of infiltrate, cavitation, or consolidation on chest x-ray obtained during the screening/baseline evaluation.
5. Use of any investigational drug or treatment up to 4 weeks prior to transplantation.
6. Treatment with voriconazole, ketoconazole, itraconazole, fluconazole, clotrimazole, astemizole, pimozide, terfenadine, erythromycin, clarithromycin, telithromycin, troleandomycin, rifampin, rifabutin, or St. John's Wort that is not discontinued prior to randomization.
7. Treatment with aminoglycosides, amphotericin B, cisplatin, cisapride, metoclopramide, cimetidine, bromocriptine, danazol, or other drugs associated with renal dysfunction that are not discontinued prior to randomization.
8. Subjects with a screening/baseline total white blood cell count < 2,000/mm3 or absolute neutrophil count (ANC) < 500, platelet count < 100,000/mm3.
9. Fasting triglycerides > 400 mg/dL (> 4.6 mmol/L) or fasting total cholesterol > 300 mg/dL (> 7.8 mmol/L) despite optimal lipid-lowering therapy.
10. History of malignancy within 2 years of enrollment (except for adequately treated basal cell or squamous cell carcinoma of the skin).
11. Auto-immune diseases inactive immunosuppressive treatment ( 3 months prior to inclusion).
12. Patient with psychiatric disorders that could be non-compliance for the treatment.
13. Non Caucasian patients.
14. Active peptic ulcers that could produce intestinal absorption disorders.
15. Subjects who are known to be human immunodeficiency virus(HIV) or hepatitis B virus (HBV) positive. Patients with hepatitis C virus (HCV) positive should be excluded if polymerase chain reaction (PCR) positive or transaminates values are ≥2 upper normal value (UNV).
16. Diabetic patients.
17. Body mass index higher than 30 Kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-03; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Percentage of biopsy-confirmed acute rejection episodes | 6 months
  To describe cumulative biopsy-confirmed acute rejection in both groups by intention to treat analysis.

SECONDARY OUTCOMES:
Percentage of steroid-sensitive acute rejection episodes | 6 months
  To describe the percentage of steroid-sensitive acute rejections rejection in both groups by intention to treat analysis.
Percentage of acute rejection episodes requiring treatment with antilymphocyte antibodies. | 6 months
  To describe the need for antibody treatment in acute rejection episodes in both groups by intention to treat analysis.
Renal function estimated by Modification of Diet in Renal Disease (MDRD) formula. | 12 months
  To describe renal function measured by MDRD in both groups by intention to treat and "on therapy" analysis.
Proteinuria measured in g/day | 6 months
  To describe proteinuria in g/day in both groups by intention to treat analysis.
Histology at month 6 protocol kidney allograft biopsy | 6 months
  To describe histology at month 6 in both groups by intention to treat and "on therapy" analysis.
Percentage of patients with negative ELISPOT | 6 months
  To describe percentage of patients with negative ELISPOT in both groups by intention to treat and "on therapy" analysis.
Percentage of patients in group A requiring CNI introduction. | 24 months
  To describe the percentage of patients in group A requiring CNI introduction.
Percentage of patients presenting adverse events requiring study withdrawal | 24 months
  To describe adverse events in the whole group ("screening failure" plus "intention to treat") in both treatments groups.
Percentage of biopsy-confirmed acute rejection episodes | 12 months
  To describe cumulative biopsy-confirmed acute rejection in both groups by intention to treat analysis.
Percentage of steroid-sensitive acute rejections rejection episodes | 12 months
  To describe the percentage of steroid-sensitive acute rejections rejection in both groups by intention to treat analysis.
Percentage of acute rejection episodes requiring treatment with antilymphocyte antibodies | 12 months
  To describe the need for antibody treatment in acute rejection episodes in both groups by intention to treat analysis.
Proteinuria measured in g/day | 12 months
  To describe proteinuria in g/day in both groups by intention to treat analysis.
Percentage of patients with negative ELISPOT | 12 months
  To describe percentage of patients with negative ELISPOT in both groups by intention to treat and "on therapy" analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Grinyó, PhD MD, Principal Investigator — Nephrology Department. Hospital de Bellvitge. Spain
Locations (2):
- Spain (2):
  - Nephrology Department. Hospital Vall d'Hebró, Barcelona, Barcelona
  - Nephrology Department. Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelone

REFERENCES:
- [Background] Bestard O, Cruzado JM, Mestre M, Caldes A, Bas J, Carrera M, Torras J, Rama I, Moreso F, Seron D, Grinyo JM. Achieving donor-specific hyporesponsiveness is associated with FOXP3+ regulatory T cell recruitment in human renal allograft infiltrates. J Immunol. 2007 Oct 1;179(7):4901-9. doi: 10.4049/jimmunol.179.7.4901. PMID 17878390
- [Background] Bestard O, Crespo E, Stein M, Lucia M, Roelen DL, de Vaal YJ, Hernandez-Fuentes MP, Chatenoud L, Wood KJ, Claas FH, Cruzado JM, Grinyo JM, Volk HD, Reinke P. Cross-validation of IFN-gamma Elispot assay for measuring alloreactive memory/effector T cell responses in renal transplant recipients. Am J Transplant. 2013 Jul;13(7):1880-90. doi: 10.1111/ajt.12285. Epub 2013 Jun 13. PMID 23763435
- [Result] Bestard O, Cruzado JM, Lucia M, Crespo E, Casis L, Sawitzki B, Vogt K, Cantarell C, Torras J, Melilli E, Mast R, Martinez-Castelao A, Goma M, Reinke P, Volk HD, Grinyo JM. Prospective assessment of antidonor cellular alloreactivity is a tool for guidance of immunosuppression in kidney transplantation. Kidney Int. 2013 Dec;84(6):1226-36. doi: 10.1038/ki.2013.236. Epub 2013 Jun 19. PMID 23783240
- See also: This is the center in Spain for the central contact and the main location including patients. — http://www.bellvitgehospital.cat/